CLINICAL TRIAL: NCT04684355
Title: Quality of Life of Colorectal Cancer Screenees in the Period Between Colonoscopy and Next Clinic Visit for Final Report: Does Real-time Endoscopic Optical Diagnosis Improve Their Quality of Life
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fu Jen Catholic University (Other)
Collaborators: Fu Jen Catholic University Hospital (Other)
Responsible Party: Principal Investigator, Chen-Ya Kuo, Attending Physician, M.D., Fu Jen Catholic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FJUH109047
Record Dates: First submitted 2020-12-21; First posted 2020-12-24 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Colorectal Neoplasms; Colonoscopy; Quality of Life; Mass Screening; Anxiety
Keywords: Colorectal Neoplasms; Colonoscopy; Quality of Life; Mass Screening; Anxiety
MeSH Terms: conditions — Colorectal Neoplasms; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard-of-care group (No Intervention): Participants in this group received their colonoscopic and pathological diagnosis simultaneously at next clinical visit, which arranged in 1 to 2 weeks later.
- Intervention group (Experimental): Participants in this group received their colonoscopic diagnosis right after they awake from general anesthesia, and then received pathological diagnosis at next clinical visit, which arranged in 1 to 2 weeks later.
  Interventions: Other: Real-time colonoscopic optical diagnosis for colorectal neoplasm

INTERVENTIONS:
Other: Real-time colonoscopic optical diagnosis for colorectal neoplasm — Colonoscopic optical diagnosis by image enhanced technology has been validated as an excellent tool to predict the histology of colorectal polyps and to differentiate the invasion depth of colorectal cancer.
  Arms: Intervention group

SUMMARY:
Colorectal cancer screening program has been proven to reduce colorectal cancer (CRC) mortality and is cost-effective. It has been adopted by most countries in the world, and colonoscopy is regarded as the most accurate test for detecting colorectal neoplasm. After screenees underwent colonoscopy, most endoscopists do not routinely explain the preliminary optical diagnosis to the subjects before they going home, which may cause unnecessary anxiety and may reduce the quality of life of the subjects before acquiring the final results. In recent years, endoscopic optical diagnostic technology has been validated by meta-analysis studies as an excellent tool to predict the histology of colorectal polyps and to differentiate the invasion depth of colorectal cancer. The real time feature of endoscopic optical diagnosis allows endoscopists to explain the preliminary results confidently to the subjects immediately after colonoscopy, which is expected to reduce the anxiety of the subjects before they acquired the final results and improve their quality of life. We designed a randomized controlled trial to validate whether real-time endoscopic optical diagnosis could decrease the anxiety burden and improve the quality of life for colorectal-cancer screenees after colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who preparing to received screening or surveillance colonoscopy under general anesthesia.
* Patients who preparing to received sedated colonoscopy due to other GI tract related symptoms.

Exclusion Criteria:

* Impaired mental status that could not understand the questionnaire questions.
* Patients with major psychological disorders.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-12-22 (Estimated); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Quality of life degree | 2 weeks
  Use WHOQOL-BREF Taiwanese version to measure the quality of life between the two study arms.

SECONDARY OUTCOMES:
Anxiety and depression degree | 2 weeks
  Use Hospital Anxiety and Depression Scale (HADS) Taiwanese version to measure the anxiety and depression degree between the two study arms.

CONTACTS AND LOCATIONS:
Locations (1):
- Fu Jen Catholic University Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No